CLINICAL TRIAL: NCT04648839
Title: Observational Retrospective Study to Characterise and Assess Clinical Outcomes of Patients Receiving Benralizumab After Marketing Approval in Spain.
Brief Title: Observational Retrospective Study on Clinical Outcomes of Patients Receiving Benralizumab in Spain.
Acronym: ORBE-II
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00079
Record Dates: First submitted 2020-10-05; First posted 2020-12-02 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Benralizumab: Patients that received at least one dose of benralizumab according to routine clinical practice

SUMMARY:
Primary Objectives:

1. To describe the demographic and baseline characteristics in patients with severe eosinophilic asthma in Spain who received at least one dose of Benralizumab, after its marketing authorization
2. To describe background treatment patterns of severe eosinophilic asthma patients at baseline and after the index date (benralizumab initiation)

This is a descriptive, observational, multi-centre, longitudinal, retrospective cohort study in adults patients (≥18 years) with severe asthma (maintenance treatment with high dose inhaled corticosteroids combined with long-acting agonist β2) and eosinophilic phenotype, who, at the discretion of the physician, received benralizumab accordingly to the clinical practice, in the period after the marketing authorization of benralizumab in Spain, on January 1st 2019.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years)
* Diagnosis of severe eosinophilic asthma requiring stable treatment of high doses of inhaled corticosteroids and a long-acting agonist β2 ± additional asthma controller.
* Patients with at least 12-month data available before index date (starting benralizumab treatment)
* Patients with at least 3-month electronic medical records data available from first benralizumab dose ("index date")
* Informed consent signed.

Exclusion Criteria:

* Patients who received benralizumab in a clinicaltrial, during the observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will be all patients with severe eosinophilic asthma (those requiring stable treatment with high doses of inhaled corticosteroids and a long-acting agonist β2 ± additional asthma controller), who received at least one dose of benralizumab according to routine clinical practice, after marketing approval on January 1st, 2019. The targeted patients need to have available medical record of 12 months prior to index date.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Age | Up to 12 months (Baseline period)
  Specifically, at the time of taking the first dose of study drug
Gender | Up to 12 months (Baseline period)
  Specifically, at the time of taking the first dose of study drug
Smoking Habits | Up to 12 months (Baseline period)
Age at athma diagnosis | Up to 12 months (Baseline period)
Blood eosinophils count | Baseline period
Total IgE | Baseline period
Number of patients with positive Prick test | Baseline period
FeNo | Baseline period
Lung function (FEV1 and FVC) | Baseline period
ACT (or ACQ) score | Baseline period
  Asthma Control Test (ACT), the scores range from 5 to 25, with higher scores reflecting greater asthma control.
  Asthma Control Questionnaire (ACQ), the total score range between 0 (well controlled asthma) and 6 (extremely poorly controlled)
AQLQ score | Baseline period
  Asthma Quality of Life Questionnaire (AQLQ), it scores from 1 (minimum) to 7 (maximum) where the higher the score, the better the quality of life is
Severe asthma exacerbations | In the previous 12 months
Key comorbidities | Baseline period
OCS-related comorbidities | Baseline period
Concomitant asthma medications | Baseline period
Physician office visits | Baseline period
  Split by primary care and specialist (asthma related)
Emergency room visits | Baseline period
Hospitalisations | Baseline period
  Number and duration
Number of laboratory tests per patient | Baseline period
Number of conventional radiology procedures per patient | Baseline period
Number of diagnostic/therapeutic tests per patient | Baseline period
  Asthma related only
Number of spirometries per patient | Baseline period
Number of allergy tests per patient | Baseline period
Number of computed axial tomographies per patient | Baseline period
Number of magnetic resonance imaging procedures per patient | Baseline period
Asthma treatment | Up to 24 months (study duration)
  Including previous biologic treatment, type of treatment and reasons for discontinuation or switching

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Madrid, Spain

REFERENCES:
- [Derived] Padilla-Galo A, Moya Carmona I, Ausin P, Carazo Fernandez L, Garcia-Moguel I, Velasco-Garrido JL, Andujar-Espinosa R, Casas-Maldonado F, Martinez-Moragon E, Martinez Rivera C, Vera Solsona E, Sanchez-Toril Lopez F, Trisan Alonso A, Blanco Aparicio M, Valverde-Monge M, Valencia Azcona B, Palop Cervera M, Nuevo J, Sanchez Tena J, Resler G, Luzon E, Levy Naon A. Achieving clinical outcomes with benralizumab in severe eosinophilic asthma patients in a real-world setting: orbe II study. Respir Res. 2023 Sep 28;24(1):235. doi: 10.1186/s12931-023-02539-7. PMID 37770889
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00079&attachmentIdentifier=8915a118-f871-450d-99d1-01c9859f044e&fileName=ORBE_II_(D3250R00079)_Study_Report_Synopsis.pdf&versionIdentifier=